CLINICAL TRIAL: NCT04544826
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of JNJ-77474462 (Bermekimab) in Healthy Participants of Japanese Descent Following Administration of Single Ascending Subcutaneous Doses
Brief Title: A Study of JNJ-77474462 (Bermekimab) in Healthy Participants of Japanese Descent Following Administration of Single Ascending Subcutaneous Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108807; 77474462ADM1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-09; First posted 2020-09-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — bermekimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: JNJ-77474462 (Low Dose) or Placebo (Experimental): Participants will receive single low dose of JNJ-77474462 or matching placebo as subcutaneous (SC) injection.
  Interventions: Drug: JNJ-77474462; Drug: Placebo
- Cohort 2: JNJ-77474462 (Medium Dose) or Placebo (Experimental): Participants will receive single medium dose of JNJ-77474462 or matching placebo as SC injection.
  Interventions: Drug: JNJ-77474462; Drug: Placebo
- Cohort 3: JNJ-77474462 (High Dose) or Placebo (Experimental): Participants will receive single high dose of JNJ-77474462 or matching placebo as SC injection.
  Interventions: Drug: JNJ-77474462; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77474462 — JNJ-77474462 will be administered as SC injection.
  Other Names: Bermekimab
Drug: Placebo — Matching placebo to JNJ-77474462 will be administered as SC injection.

SUMMARY:
The purpose of the study is to assess the safety and tolerability of JNJ-77474462 following single subcutaneous (SC) administration to healthy participants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be of first to third generation Japanese descent
* Participant must be otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and Day-1. Any abnormalities, must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be otherwise healthy on the basis of clinical laboratory tests performed at screening and Day-1. If the results of the serum chemistry panel including hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) (BMI = weight/height^2) and a body weight of between 50 to 90 kg inclusive
* A female participant must have a negative pregnancy test at screening and on Day -1

Exclusion Criteria:

* Coexisting Medical Conditions or Past Medical History: History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, endocrine, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Coexisting Medical Conditions or Past Medical History: Has known allergies, hypersensitivity, or intolerance to JNJ-77474462 or its excipients, or any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies or antibody fragments, or to any components of the formulation of JNJ-77474462 and its excipients used in this study
* Malignancy or Increased Potential for Malignancy: Has a history of malignancy before screening. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk and no evidence of recurrence within 5 years prior to screening
* Concomitant or Previous Medical Therapies Received: Participant is currently enrolled in an investigational study or has received an investigational intervention (including investigational vaccines or devices) 5 half-lives or 8 weeks prior to screening (whichever is longer)
* Concomitant or Previous Medical Therapies Received: Has received over the counter medications (including vitamins/multivitamins supplements, corticosteroids, acetaminophen/paracetamol, aspirin, decongestants, antihistamines and other non-steroidal anti-inflammatory drugs), and herbal medication (including, but not limited to, herbal tea, St. John's Wort, and cannabidol) within 2 weeks prior to first study intervention administration unless approved by the investigator and sponsor medical monitor
* Infections or Predisposition to Infections: has an active acute or clinically significant chronic infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Week 16
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 16
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) by System Organ Class (SOC) Reported in two or More Participants | Up to Week 16
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Week 12
  Number of participants with clinically significant changes in vital signs (temperature, pulse/heart rate, respiratory rate, blood pressure) will be reported.
Number of Participants with Clinically Significant Changes in Electrocardiograms (ECGs) Waveform | Up to Week 12
  Number of participants with clinically significant changes in ECGs waveform (example: changes in T-wave morphology or the occurrence of U-waves) will be reported.
Number of Participants with Clinically Significant Changes in Hematology | Up to Week 12
  Number of participants with clinically significant changes in hematology (such as platelet count, Red blood cell count [RBS], Hemoglobin, Hematocrit, RBC Indices, WBCs) will be reported.
Number of Participants with Clinically Significant Changes in Chemistry | Up to Week 12
  Number of participants with clinically significant changes in chemistry (such as Sodium, Potassium, Chloride, Bicarbonate,glucose, Total bilirubin, Uric acid) will be reported.
Number of Participants with Clinically Significant Changes in Urinalysis | Up to Week 12
  Number of participants with clinically significant changes in urinalysis (such as Specific gravity, pH, Glucose,Protein, WBCs, Bacteria) will be reported.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Up to Week 12
  Cmax is the maximum observed concentration.
Area Under the Plasma/Serum Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) | Up to Week 12
  AUC(0-infinity) is defined area under the plasma/serum concentration versus time curve from time zero to infinity with extrapolation of the terminal phase.
Area Under the Plasma/Serum Concentration-time Curve from Time Zero To Time Of the Last Quantifiable Concentrations (AUC[0-last]) | Up to Week 12
  AUC(0-last) is defined as area under the plasma/serum concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Time to Reach Maximum Observed Concentration (Tmax) | Up to Week 12
  Tmax is the time to reach maximum observed concentration.
Terminal Half-life (T1/2) | Up to Week 12
  T1/2 is the terminal half-life.
Apparent Total Systemic Clearance (CL/F) | Up to Week 12
  CL/F is the apparent total systemic clearance after extravascular administration.
Apparent Volume of Distribution (Vz/F) | Up to Week 12
  Vz/F is the apparent volume of distribution based on terminal phase after extravascular administration.
Number of Participants with Antibodies to JNJ-77474462 | Up to Week 12
  Number of participants with antibodies to JNJ-77474462 in participants receiving active study active intervention in total and by intervention group will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Nucleus Network, Q-Pharm Pty Ltd, Herston, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency